CLINICAL TRIAL: NCT05803291
Title: Children With Special Health Needs. Evaluation of Continuity of Care and Integrated Hospital-territory Care Pathways in Friuli Venezia Giulia
Brief Title: Evaluation of Continuity of Care of Children With Special Health Needs
Status: Completed | Type: Observational
Sponsor: IRCCS Burlo Garofolo (Other)
Responsible Party: Sponsor
Other Study IDs: RC 17/16
Record Dates: First submitted 2023-03-24; First posted 2023-04-07 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Children With Special Health Needs
Keywords: Special health needs; Continuity of care; Care coordination; Children

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Children and adolescents with special health care needs represent a small but relevant subset of the pediatric population due to high costs for the health care system, risk of lower quality of care, unmet health care needs, and negative health outcomes. Coordination of care and continuity of care are essential issues of appropriate care for these patients, as showed also by the "Special Needs Kids" project, carried out in Emilia Romagna. This project showed the potential for family pediatricians (FP) in Italy to serve as care coordinators and facilitate the implementation of integrated care pathways for children with special health care needs. In Friuli-Venezia Giulia (FVG), a system of "continuity of care" for patients with special needs was developed and implemented. This system integrate hospital and community care in a network involving also FPs, General Practitioner and different actors of social and health services. The aim of this study is to prospectively evaluate the continuity of care provided to children and adolescents with special health needs residing in the FVG region.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with special health care needs requiring continuity of care and integrated home care
* Age between 0 to 17 years
* Residence in FVG region
* Outpatient, inpatient or emergency care admission at the IRCCS Burlo Garofolo hospital, Trieste, Italy

Exclusion Criteria:

-

Ages: 1 Day to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study involves pediatric patients with special health care needs recruited at IRCCS Burlo Garofolo over a 12-month period and followed prospectively for the next 12 months (follow-up)
Sampling Method: Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2018-09-26 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
To assess health care providers activities using the Special Needs Kids instrument | Through study completion, an average of 12 months
  The Special Needs Kids (SpeNK)-FP instrument includes eight descriptive items aiming to collect information about the activity performed by the FP for the patients, involving the child or the family and including visit at the clinic, phone contact, ecc. In particular, SpeNK-FP evaluates: patient's clinical and social complexity on a three levels scale; requests or problems addressed; needs for care coordination; activities carried out by the FP; involvement of any other professionals in the care coordination activity; time spent for care coordination; FP's appraisal about the outcomes occurred and prevented with the care coordination activity.
To assess parents' perspective on continuity of care using the Special Needs Kids Questionnaire | At 10 months after enrollment
  The Special Needs Kids Questionnaire (SpeNK-Q) is a 20 items (with 5-point response option) questionnaire, evaluating parents' perspective about their relationship and interactions with: 1) the FP; 2) the main care coordinator; 3) the network of health care providers and services. SpeNK-Q includes two open questions aiming at identifying: 1) the person who is in charge of most of the child's health; (2) the person who coordinates the child's health care. The 5-point response option are: from "fully disagree" to "fully agree" for questions 1-7 concerning FP (lower scores indicates a worse outcome); form "never or almost never" to "always or almost always" for questions 8-20 concerning the network of health care providers and services.

CONTACTS AND LOCATIONS:
Overall Officials: Elisa Zanello, MSC, Principal Investigator — IRCCS materno infantile Burlo Garofolo
Locations (1):
- IRCCS Burlo Garofolo, Trieste, Italy